CLINICAL TRIAL: NCT02935400
Title: Acute Porphyrias: Biomarkers for Disease Activity and Response to Treatment
Brief Title: Acute Porphyria Biomarkers for Disease Activity
Status: Active, not recruiting | Type: Observational
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Other Study IDs: 14-0001
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Acute Intermittent Porphyria; Hereditary Coproporphyria; Variegate Porphyria
Keywords: porphyria; biomarkers
MeSH Terms: conditions — Porphyria, Acute Intermittent; Coproporphyria, Hereditary; Porphyria, Variegate; Porphyrias | interventions — Hemin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 1. Blood specimens collected in Paxgene tubes for isolation of RNA for expression studies.
  2. Blood samples for metabolomic studies
  3. Urine samples for metabolomic studies
  4. Stool samples for metabolomic studies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Asymptomatic: Group 1 will have had no symptoms of porphyria in the past year.
- Symptomatic and treated with hemin: Group 2 will have a history of symptoms within the past year.
  Interventions: Drug: Hemin

INTERVENTIONS:
Drug: Hemin — Hemin will be administered under a separate protocol or for clinical treatment, and samples will be collected under this protocol before and after treatment.
  Other Names: Panhematin
  Groups: Symptomatic and treated with hemin

SUMMARY:
The long term objective of the research is to identify new biomarkers of disease activity in the human acute porphyrias. This pilot study is intended to provide pilot and feasibility data needed to plan larger and more definitive future studies.

DETAILED DESCRIPTION:
This translational pilot research is based on preliminary results using animal models. The investigators will collect samples of blood, urine and feces from up to 50 participants with well documented acute porphyrias, at 2 expert sites that are members of the Porphyrias Consortium. Collection and analysis of these samples will be used to assess feasibility of performing such studies in humans with acute porphyrias, recognizing that these disorders are more heterogeneous than reproduced in animal models, and affect individuals who cannot all be studied simultaneously and in large groups. Therefore, we will assess the feasibility of methods for collecting, processing, storing and shipping samples at multiple study sites for later biomarker analysis. Larger and more definitive studies of biomarkers will be designed and implemented based on data and experience from this pilot-feasibility study.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of acute porphyria.

  1. For AIP: Elevation in urine PBG, with normal or only slight increases in plasma and fecal porphyrins. Most (~90%) will have deficient activity of erythrocyte PBGD.
  2. For HCP: Elevation in urine PBG, with substantial increases in fecal porphyrins (almost entirely coproporphyrin III). In the absence of skin photosensitivity, most will have normal or only slight increases in plasma porphyrins.
  3. For VP: Elevation in PBG, with substantial increases in fecal porphyrins (mostly coproporphyrin III and protoporphyrin), increased plasma total porphyrins and a fluorescence emission maximum of diluted plasma at neutral pH near 626 nm.

Exclusion Criteria:

* Another medical condition that might confound the results, as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute intermittent porphyria, hereditary coproporphyria, variegate porphyria.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-04-28 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Potential biomarkers Biomarkers | 10 days
  Expression of heme biosynthetic and heat and stress response genes

CONTACTS AND LOCATIONS:
Overall Officials: Karl E Anderson, Principal Investigator — University of Texas
Locations (1):
- University of Texas Medical Branch, Galveston, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data not entered